CLINICAL TRIAL: NCT06884306
Title: Predictors of Spontaneous Bacterial Peritonitis Among Patients with Cirrhosis
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Nashaat Mohamed Ahmed, residant doctor, Assiut University
Other Study IDs: SBP Cirrhosis
Record Dates: First submitted 2025-03-13; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- study group: cirrhotic patients with Moderate-marked ascites, as determined by abdominal ultrasonography (US). SBP will be diagnosed based on detection of polymorph nuclear leukocytes (PMNs) >250 cells/mcL and/or white blood cells (WBCs) >500 cells/mcL by ascitic fluid examination.

SUMMARY:
Prevalence of spontaneous bacterial peritonitis (SBP) varies from approximately 4% among asymptomatic patients to 30% among those hospitalized [1, 2].Previous studies explored the role of several biomarkers, such as tumor necrosis factor-α, procalcitonin, and fecal calprotectin, for prediction of SBP The NLR is speculated to reflect immune regulatory mechanism (lymphocytes) and ongoing inflammation (neutrophils) . Assessing the diagnostic value of NLR for liver disease has gained particular interest, namely, among patients with nonalcoholic fatty liver disease and hepatocellular carcinoma . Direct interaction between platelets and bacteria lead to platelet activation . Platelet activation leads to change of platelet shape with increase in platelet size and anisocytosis, and consequent increase in both mean platelet volume (MPV) and platelet distribution width (PDW) .Acute phase reactants, such as C-reactive protein (CRP) and erythrocyte sedimentation rate (ESR), are elevated among patients with SBP, as a result of cytokine synthesis . Older patients, due to higher possibility of advanced liver disease and more frequent comorbidity, are more susceptible to SBP .

The Department of Tropical Medicine (Mansoura University) developed a simple scoring system for prediction of SBP among cirrhotic patients with ascites, which include four variables: age, MPV, NLR, and C-reactive protein (CRP) . The independent predictors of SBP were age of at least 55 years, MPV of at least 8.5 fL, NLR of at least 2.5, and CRP of at least 40 mg/dL . The progression of hospitalized patients with SBP can lead to an in-hospital mortality rate of approximately 17% .

Therefore, the sequelae of SBP highlight the increasing value of establishing reliable diagnostic biomarkers. The earlier the diagnosis, the lower the mortality rate.To our knowledge, only one, national study utilized MPV, NLR, and CRP for prediction of SBP among cirrhotic patients with ascites [3].We intend to further extend both the diagnostic utilities (by adding ESR to the previously mentioned tools) and the spectrum of prediction, to include mortality in addition to the development of SBP among cirrhotic patients with ascites.

The study aims at developing a local scoring system (RSS) for the prediction of SBP and its related mortality among cirrhotic patients with ascites admitted to Al-Rajhy Liver Hospital (Assiut University).

Our objective is to compare age, NLR, MPV, PDW, and CRP between cirrhotic patients with ascites complicated with SBP and those without SBP, and between surviving SBP patients compared to those with in-hospital mortality.

ELIGIBILITY:
Inclusion Criteria:

* include cirrhotic patients with Moderate-marked ascites, as determined by abdominal ultrasonography (US). SBP will be diagnosed based on detection of polymorph nuclear leukocytes (PMNs) >250 cells/mcL and/or white blood cells (WBCs) >500 cells/mcL by ascitic fluid examination.

Exclusion Criteria:

* 1- Pediatric patients (less than 18 years old) and patients older than 70 years Pregnant patients .

  2-Etiology of ascites other than cirrhosis. 3-Receiving antibiotics and/or prophylaxis four weeks before admission. 4- Concurrent bacterial infection other than SBP. 5- Abdominal surgery 12 weeks before admission 6-Patients with neoplastic or hematological disease. 7- Patients who received bone marrow transplantation, chemotherapy, or radiotherapy four weeks before admission.

  8- Conditions associated with increased MPV such as systemic hypertension, diabetes mellitus, dyslipidemia, peripheral vascular disease, thyroid disease, and therapy four weeks before admission with antiplatelet agents and nonsteroidal anti-inflammatory drugs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cirrhotic patients with Moderate-marked ascites, as determined by abdominal ultrasonography (US). SBP will be diagnosed based on detection of polymorph nuclear leukocytes (PMNs) >250 cells/mcL and/or white blood cells (WBCs) >500 cells/mcL by ascitic fluid examination.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
local scoring system (RSS) | baseline
  developing a local scoring system (RSS) for the prediction of SBP mortality among cirrhotic patients with ascites admitted to Al-Rajhy Liver Hospital (Assiut University